CLINICAL TRIAL: NCT06034015
Title: A Phase 1, Two-Part, Open-Label Study to Evaluate the Safety, Tolerability and Pharmacokinetics (PK) of Single Ascending Doses of APL-1501 Extended Release (ER) Capsules Compared to APL-1202 Immediate Release (IR) Tablets in Healthy Volunteers (Part A) and Multiple Ascending Doses of APL-1501 ER Capsules Compared to APL-1202 IR Tablets in Healthy Volunteers (Part B)
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of APL-1501 Extended Release (ER) Capsules Compared to APL-1202 Immediate Release (IR) Tablets in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YHGT-PN-02
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Active Comparator)
  Interventions: Drug: APL-1202 and APL-1501 (Single ascending dose)
- Part B (Active Comparator)
  Interventions: Drug: APL-1202 and APL-1501 (Multiple Ascending dose)

INTERVENTIONS:
Drug: APL-1202 and APL-1501 (Single ascending dose) — Period 1 drug adminstration (APL-1202 IR tablet , single dose of 375mg will be administered orally on Day 1; washout period of 72 hrs; Period 2 drug administration (APL-1501 ER capsules of 764mg, 1146 mg and 1528 mg will be administered as single dose on Day 4.
  Arms: Part A
Drug: APL-1202 and APL-1501 (Multiple Ascending dose) — Period 1 drug adminstration (APL-1202 IR of 375mg will be administered thrice a day (TID) orally from Day 1 to Day 5; washout period of 72 hrs; Period 2 drug administration (APL-1501 ER capsules of 764mg, 1146 mg and 1528 mg will be administered twice daily (BID) from Day 9 to 13.
  Arms: Part B

SUMMARY:
This is an integrated Phase 1, single centre, 2-part, open-label, dose-escalation study conducted in healthy volunteers to assess the safety, tolerability, and PK of APL-1501 ER capsules in comparison to APL-1202 IR tablets.

DETAILED DESCRIPTION:
The study will have 2 parts: Each study part will comprise 2 dosing periods with a 72-hour washout period in between:

Period 1: APL-1202 IR tablet dosing and Period 2: APL-1501 ER capsule dosing.

In Part A dosing will be single day/single dosing for the APL-1202 IR tablets, and single day/single dosing the APL-1501 ER capsules with 24 participants in 3 sequential cohorts, Cohorts A1, A2, and A3. Each cohort will enrol 8 participants, with male to female participants in a 1:1 ratio. In Period 1/Day 1, participants in all cohorts will be dosed with single dose of 375 mg APL-1202 IR tablets which will followed by a washout period of at least 72 hours, after which participants will be dosed with single dose of APL-1501 ER capsules in Period 2/Day 4, .

In Part B dosing will be multi-day/TID dosing for the APL-1202 IR tablets, and multi-day/BID dosing the APL-1501 ER capsules with 24 participants in 2 sequential cohorts, Cohorts B1 and B2. Each cohort will enrol 12 participants, with male to female participants in a 1:1 ratio and in each of the 2 study periods, participants will be administered IP for 5 days. In period 1, participants will administered with APL-1202 IR tablet (TID) on Day 1, Day 2, Day 3, Day 4, and Day 5 and period 2 with APL-1501 ER capsule (BID) dosing on Day 9, Day 10, Day 11, Day 12, and morning of Day 13.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female 18 to 65 years of age (inclusive at the time of informed consent).
2. In good general health, with no significant medical history and no clinically significant abnormalities on physical examination, 12-lead ECG, vital signs and oximetry measurements at Screening and/or before the first administration of Investigational Products (IP), as determined by the Principal Investigator or designee.
3. Clinical laboratory values within normal range as specified by the testing laboratory, at Screening and/or before the first administration of IP unless deemed not clinically significant (NCS) by the Principal Investigator or designee.
4. Body-mass index (BMI) between ≥ 18.0 and ≤ 32.0 kg/m2 at Screening and weight ≥ 50 kg.
5. Current non-smoker or casual smoker who used no more than 5 cigarettes (or equivalent quantity of any other nicotine-containing products eg, snuff, chewing tobacco, cigars, cigarettes, pipes, e-cigarettes [Vaping] etc.) per week for 3 months prior to Screening. Participants must abstain from smoking and abstain from using nicotine-containing products (eg, nicotine chewing gum, nicotine plasters, or other product used for smoking cessation) for 2 weeks prior to admission and throughout the study period, and test negative at Screening and on Day -1 for urinary cotinine.
6. No relevant dietary restrictions.
7. Females must not be pregnant or lactating, and must use acceptable, highly effective double contraception from Screening until 30 days after study completion, including the Follow-up period.
8. Males must be surgically sterile (> 90 days since vasectomy with no viable sperm), or if engaged in sexual relations with a women of child bearing potential (WOCBP), his partner must be either surgically sterile (eg, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or use an acceptable, highly effective contraceptive method (see Section 7.3.3) from Screening until 90 days after study completion, including the Follow-up period.
9. Able and willing to attend the necessary visits to the study site.
10. Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

1. Underlying physical or psychological medical condition that, in the opinion of the PI, would make it unlikely for the participant to comply with the protocol or complete the study per protocol.
2. Receipt of blood products, or significant blood loss deemed to be CTCAE Grade 3 or Grade 4 within 6 weeks prior to the first administration of IP.
3. Plasma donation within 7 days prior to the first administration of IP, or platelet/blood donation within 4 weeks prior to the first administration of IP
4. Fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to the first administration of IP.
5. Poor pill swallowing ability.
6. History of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents, including lactose intolerance/allergy.
7. History of malignancy, except for non-melanoma skin cancer, excised more than 1 year prior to Screening and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
8. History or presence of a condition associated with significant immunosuppression.
9. History of life-threatening infection (eg, meningitis). Severe infections within 4 weeks prior to the first administration of IP including but not limited to hospitalisation for complications of infection, bacteraemia, or severe pneumonia.
10. Infections requiring parenteral antibiotics within 6 months prior to the first administration of IP.
11. Vaccination with a live vaccine within 4 weeks prior to the first administration of IP. COVID-19 or influenza can be exempted.
12. Exposure to any significantly immune suppressing drug (including experimental therapies as part of a clinical study) within 4 months prior to the first administration of IP or 5-half-lives, whichever is longer.
13. Positive test for hepatitis C virus antibody (HCVAb), hepatitis B virus surface antigen (HBsAg), human Immunodeficiency virus (HIV) antibody, or COVID-19 at Screening and Day-1.
14. History of tuberculosis (TB) or positive QuantiFERON®-TB Gold test at Screening or 2 successive indeterminate QuantiFERON-TB Gold test results.
15. Positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol, amphetamines, benzodiazepines, opiates, cocaine and tricyclic antidepressants), or alcohol breath test at Screening and Day-1.
16. History of substance abuse or dependency or history of recreational intravenous drug use over the last 5 years (by self-declaration).
17. Regular alcohol consumption defined as > 10 standard drinks per week (where 1 standard drink = 360 mL of beer, 45 mL of 40% spirit or a 150 mL glass of wine) or > 4 standard drinks on any single day. Participant is unwilling to abstain from alcohol beginning 48 hours prior to the first administration of IP and for the duration of the study.
18. Use of any IP or investigational medical device within 30 days prior to the first administration of IP, or 5 half-lives of the product (whichever is the longest), or participation in more than 4 investigational drug studies within 1 year prior to the first administration of IP.
19. Use of (or anticipated use of) any prescription drugs or over-the-counter (OTC) medication, herbal remedies, supplements or vitamins 2 weeks prior to the first administration of IP and during the course of the study without prior approval of the PI and Medical Monitor (MM). Simple analgesia (paracetamol, nonsteroidal anti-inflammatory drug ) may be permitted at the discretion of the PI. The use of hormonal contraception, oral contraceptive pills, long-acting implantable hormones, injectable hormones, a vaginal ring, or an intrauterine device (IUD) will be permitted.
20. Unwilling to refrain from strenuous exercise (including weightlifting) 48 hours prior to the admission to the clinical research unit (CRU) and 48 hours prior to any outpatient visit.
21. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, ophthalmological or psychiatric disorder, as determined by the PI or designee, if deemed clinically relevant by PI or designee.
22. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs. Uncomplicated appendectomy, uncomplicated cholecystectomy and hernia repair will be allowed as determined by the PI or designee.
23. Use or intent to use any medications/products/food known to alter drug absorption, metabolism, or elimination processes, including strong inducers or inhibitors of metabolism enzymes or transporters, including but not limited to St. John's wort, grapefruit, and grapefruit juice, within 14 days prior to the first administration of IP, unless deemed acceptable by the PI or designee.
24. A participant who, in the opinion of the PI or designee, should not participate in this study
25. Anything that the PI considers would jeopardise the safety of the participant, prevent complete participation in the study, or compromise interpretation of the study data.
26. Smoked more than 5 cigarettes per week 3 months prior to Screening.
27. Has a positive cotinine at Screening and on Day -1 and or disagreed abstinence from the use of any tobacco products 2 weeks prior to admission to the CRU and throughout the study period.
28. Optic nerve disease and cataracts and those with a history of related conditions

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-09 (Estimated); Primary Completion 2024-01-19 (Estimated); Study Completion 2024-02-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Part A: upto Day 11 post dose follow up; Part B: Upto Day 20 post dose follow up
  Number of participants with AEs
Serious Adverse Events (SAEs) | Part A: upto Day 11 post dose follow up; Part B: Upto Day 20 post dose follow up
  Number of participants with SAEs
Treatement Emergent Adverse Events (TEAEs) | Part A: upto Day 11 post dose follow up; Part B: Upto Day 20 post dose follow up
  Number of participants with TEAEs

SECONDARY OUTCOMES:
PK parameters: area under the curve (AUC) | up to 120 hours post dose in each treatment period
  Area under the curve (AUC) of APL-1501 ER capsules and APL-1202 IR Tablets
PK parameters: maximum concentration (Cmax) | up to 120 hours post dose in each treatment period
  maximum concentration (Cmax), of APL-1501 ER capsules and APL-1202 IR Tablets
PK parameters: Tmax | up to 120 hours post dose in each treatment period
  Tmax of APL-1501 ER capsules and APL-1202 IR Tablets
PK parameters: half-life (t1/2) | up to 120 hours post dose in each treatment period
  apparent t1/2 of APL-1501 ER capsules and APL-1202 IR Tablets
Urine PK parameters: Renal clearance (CLr) | up to 120 hours post dose in each treatment period
  Urine concentration of APL-1202 Tablets.
Urine PK parameters: Total amount of the APL-1202 excreted in urine from time t1 to t2 hours (Aet1-t2) | up to 120 hours post dose in each treatment period
  Urine concentration of APL-1202 Tablets.
PK Parameters: Apparent total plasma clearance (CL/F) | up to 120 hours post dose in each treatment period
  CL/F of APL-1501 ER capsules and APL-1202 IR Tablets
PK Parameters: Apparent terminal volume of distribution (Vz/F) | up to 120 hours post dose in each treatment period
  Vz/F of APL-1501 ER capsules and APL-1202 IR Tablets

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No